CLINICAL TRIAL: NCT01430078
Title: A Phase 1, Open-Label, 4-Way Crossover Regional Drug Absorption Study to Assess the Bioavailability of ASP015K in Healthy Subjects
Brief Title: A Study to Assess the Bioavailability of ASP015K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 015K-CL-PK15; 2010-021160-15 (EudraCT Number)
Record Dates: First submitted 2011-06-08; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: ASP015K; Healthy subjects; Pharmacokinetics of ASP015K
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regimen A (Experimental): ASP015K oral tablet
  Interventions: Drug: ASP015K
- Regimen B (Experimental): ASP015K solution delivered to distal small bowel via oral capsule
  Interventions: Drug: ASP015K
- Regimen C (Experimental): ASP015K solution delivered to ascending colon via oral capsule
  Interventions: Drug: ASP015K
- Regimen D (Experimental): ASP015K solution delivered to distal transverse colon via oral capsule
  Interventions: Drug: ASP015K

INTERVENTIONS:
Drug: ASP015K — oral tablet
  Arms: Regimen A
Drug: ASP015K — solution via oral capsule
  Arms: Regimen B; Regimen C; Regimen D

SUMMARY:
The objective of the study is to assess the bioavailability of ASP015K within the gastrointestinal tract.

DETAILED DESCRIPTION:
Each subject will participate in four separate study periods. In each period, subjects will be admitted to the clinical unit approximately seven hours on the day prior to being given study drug. Subjects will remain at the clinical research unit for the next 24 hours after they have received study drug. Subjects will return to the clinical research unit at 36 and 48 hours after they have received study drug to give blood samples. There will be a minimum of a four day "washout" period, between each study period.

Under certain circumstances, subjects may be asked to return to the clinical research unit for an additional study period.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighing at least 45 kg and BMI of 18-32 kg/m2
* Subject must demonstrate their ability to swallow an empty size 000 capsule
* Subject agrees to sexual abstinence, is surgically sterile (with documentation provided by a healthcare professional), or is using a medically acceptable method to prevent pregnancy during the study
* Subject has a normal 12-lead ECG
* Subject is medically healthy, with no clinically significant medical history or abnormalities

Exclusion Criteria:

* Subject has ever sought advice from, or been referred to, a General Practitioner (GP) or counselor for abuse or misuse of alcohol, non medical drugs, medicinal drugs or other substance abuse e.g. solvents
* Subject is currently using or has had previous use of Class A drugs such as opiates, cocaine, ecstasy, lysergic acid diethylamide (LSD) and intravenous amphetamines
* The subject has a positive drugs of abuse test result
* The subject regularly consumes alcohol >21 units per week
* The subject is a current smoker or has smoked within the last 12 months
* The subject has clinically significant abnormal biochemistry, hematology or urinalysis
* The subject has a history of gastrointestinal surgery (with the exception of appendectomy unless it was performed within the previous 12 months)
* The subject has a history of clinically significant cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome
* The subject has had radiation exposure from clinical trials exceeding 5 mSv in the last twelve months or 10 mSv in the last five years
* The subject has a history of adverse reaction or allergy to study drug or its excipients The subject suffers from hayfever they must not have or be expecting to have symptoms during the study
* The subject has had acute diarrhoea or constipation in the 7 days before the first study day
* The subject has the presence of non-removable metal objects such as metal plates, screws, etc, in the abdominal region of the body (with the exception of sterilisation clips)
* The subject has a positive Hepatitis B virus (HBV), Hepatitis C virus (HCV) or Human Immunodeficiency virus HIV results
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to study drug administration, or over the counter medication within 7 days prior to study drug administration
* The subject has/had a symptomatic, viral, bacterial, or fungal infection within 1 week prior to clinic check in
* The subject has been vaccinated within the last 90 days
* The subject has participated in a clinical research study involving investigational drugs or dosage forms within the previous 90 days
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 90 days or donated plasma within 7 days prior to clinic admission
* The subject has a past history of tuberculosis or absence of evidence of successful TB immunization as assessed at clinical examination of the Bacille Calmette-Guérin (BCG) scar
* The subject has a past history of recurrent herpes simplex or varicella zoster infections

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment of AUC through the analysis of blood samples | Up to 45 days

SECONDARY OUTCOMES:
Pharmacokinetic assessment of maximum concentration (Cmax) through the analysis of blood samples | Up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Quotient Clinical Limited, Ruddington, Nottingham, United Kingdom